CLINICAL TRIAL: NCT05560503
Title: Establish a New Noninvasive Diagnostic Model Based on Common Clinical Indicators to Evaluate the Liver Fibrosis in Patients With Chronic Hepatitis B
Brief Title: A Nomogram for Evaluating Significant Liver Fibrosis in Patients With Chronic Hepatitis B Virus Infection
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202205120
Record Dates: First submitted 2022-08-29; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-08

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- significant liver fibrosis: According to the Scheuer scoring system, the degree of fibrosis S2-S4 as significant liver fibrosis.
- non-significant liver fibrosis: According to the Scheuer scoring system, the degree of fibrosis S0-S1 was defined as non-significant liver fibrosis.

SUMMARY:
Liver fibrosis is the key step for progression to cirrhosis and liver cancer in patients with chronic hepatitis B (CHB). It is crucial to identify significant liver fibrosis in the treatment of CHB patients. Hence, the investigators aim to construct and validate a new nomogram model for evaluating significant liver fibrosis in CHB patients. The nomogram was based on a retrospective study of 259 CHB patients, who underwent liver biopsy. Through random grouping, 182 cases (70%) were included in the training set and 77 cases (30%) were included in the validation set. Biopsy pathological stage was used as the gold standard to screen the factors included in the model. The receiver operating characteristic (ROC), area under the ROC curve (AUC), calibration curve, and decision curve analysis were used to evaluate the diagnostic effect of this nomogram model. In addition, the investigators will compare the diagnostic efficiency of the new nomogram model with APRI, FIB-4, and GPR.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic standard presented in Asian-Pacific clinical practice guidelines on the management of hepatitis B.
* HBsAg-positive for over 6 months.
* aged 18-65 years old.
* no gender limitation.

Exclusion Criteria:

* co-infection with other types of hepatitis viruses, including types A, C, D, and E.
* co-infection with human immunodeficiency virus (HIV).
* autoimmune hepatitis (AIH), primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), inherited metabolic liver disease, drug-induced liver injury (DILI), alcoholic liver disease, and hepatocellular carcinoma (HCC).
* with other malignant tumor and other major systemic diseases.
* incomplete clinical data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2017 to May 2022, a total of 259 patients with chronic hepatitis B who underwent liver biopsy, in Xiangya Hospital of Central South University, were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Differences in demographic data and clinical test indicators between significant liver fibrosis group and non-significant liver fibrosis group | 0 week
  Demographic data include age and sex. Dlinical test indicators include albumin, total bilirubin, alanine aminotransferase, aspartate aminotransferase, γ-glutamyl transferase, alkaline phosphatase, white blood cell count, neutrophil count, hemoglobin, platelet count, prothrombin activity, international normalized ratio, activated partial thromboplastin time, alpha fetoprotein, HBV DNA, HBsAg, and HBeAg.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol